CLINICAL TRIAL: NCT03866421
Title: Prevalence and Metabolic Impact of Non-alcoholic Fatty Liver Disease in Patients With Chronic Kidney Disease and the Effect of Kidney Transplantation on These Parameters
Brief Title: NAFLD Among Patients With Chronic Kidney Disease and the Effect of Kidney Transplantation
Status: Terminated | Type: Observational
Why Stopped: Due to recruitment as we were challenged in finding patients eligible for the study.
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other); Herlev and Gentofte Hospital (Other); The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Bo Feldt-Rasmussen, Professor, Head of the Department of Nephrology, Rigshospitalet, Denmark
Other Study IDs: NAFLD and CKD - Study 2
Record Dates: First submitted 2019-01-30; First posted 2019-03-07 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Chronic Kidney Diseases; PreDiabetes; Kidney Transplant
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Renal Insufficiency, Chronic; Prediabetic State | interventions — Continuous Glucose Monitoring; Glucose Tolerance Test; Absorptiometry, Photon; Blood Specimen Collection; Demography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for both immediately analyses (basic lab data) and later analyses (bile acids, glucagon, amino acids, GLP-1, GIP, lipidomics and metabolomics) and stored for 10 years whereafter they will be destroyed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Kidney transplanted patients: Number of patients: 16
  Patients on the waiting list for kidney transplantation with a living donor. The patients are screened with an OGTT before participation in the study, thereby excluding patients with diabetes mellitus.
  Patients in this group are examined three times (baseline (before transplantation) and after three and twelve months after transplantation).
  Same interventions as in the control Group.
  Including/ Exclusion criteria are listed under the section "Eligibility"
  Interventions: Diagnostic Test: MR spectroscopy of the liver; Diagnostic Test: Fibroscan of the liver; Device: Continuous glucose monitoring (CGM) for four days.; Diagnostic Test: Oral glucose tolerance test (OGTT); Diagnostic Test: Intra venous glucose infusion (IIGI); Radiation: Dual Energy X-ray Absorptiometry (DEXA) scan; Biological: Blood samples; Other: Clinical and demographic data
- Control group: Number of patients: 16
  Participants in this group are matched on age and BMI according to the kidney transplanted patients.
  Participants are screened with an OGTT before participation since only persons with normal glucose tolerance may be included in the study.
  Furthermore, participants have to have normal kidney function.
  Participants in this group are only examined once. Same interventions as in the kidney transplanted patient group
  Interventions: Diagnostic Test: MR spectroscopy of the liver; Diagnostic Test: Fibroscan of the liver; Device: Continuous glucose monitoring (CGM) for four days.; Diagnostic Test: Oral glucose tolerance test (OGTT); Diagnostic Test: Intra venous glucose infusion (IIGI); Radiation: Dual Energy X-ray Absorptiometry (DEXA) scan; Biological: Blood samples; Other: Clinical and demographic data

INTERVENTIONS:
Diagnostic Test: MR spectroscopy of the liver — Magnetic resonance spectroscopy of the liver. Golden standard for non-invasive determination of NAFLD
Diagnostic Test: Fibroscan of the liver — Transient Elastography for Measurement of liver fibrosis.
Device: Continuous glucose monitoring (CGM) for four days. — CGM is attached to the abdominal skin for four days. Afterwards data is converted and analysed in a computer program.
Diagnostic Test: Oral glucose tolerance test (OGTT) — OGTT with incretin hormones. Measured for three hours.
Diagnostic Test: Intra venous glucose infusion (IIGI) — This test is combined with the OGTT to compare responses of parenteral vs enteral stimulation. The test is followed by a bolus of 5 g of L-arginin.
Radiation: Dual Energy X-ray Absorptiometry (DEXA) scan — DEXA-scan of the body composition.
Biological: Blood samples — Immediately analyse of basic lab data. Later analyses for glucagon, amino acids, bile acids, lipidomics and metabolomics.
Other: Clinical and demographic data — Measurements of blood pressure, pulse, height, weight.

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease in developed countries affecting approximately 30 % of the general adult population. It represents an important pathogenic factor in the development of type 2-diabetes and is associated with a high risk of cardiovascular disease. Previous studies of patients with chronic kidney disease (CKD) have demonstrated an increased risk for NAFLD and the presence of both CKD and NAFLD is likely to increase the risk for cardiovascular disease.

The present protocol describes a study of the prevalence and etiology of NAFLD among patients scheduled for kidney transplantation and the possible effect of kidney transplantation on NAFLD.

The project is a prospective cohort study. The effect of kidney transplantation in patients with prediabetes or normal glucose tolerance compared to healthy controls will be examined regarding development and progression of fat accumulation in the liver.

Fat accumulation in the liver will be determined by magnetic resonance (MR) spectroscopy and the prevalence of NAFLD in the two groups will be investigated. A continuous glucose monitoring (CGM) for four days, Dual Energy X-ray Absorptiometry (DEXA) scanning, fibro scanning of the liver, bile acid analysis, metabolomic and lipidomic analysis will also be performed.

An oral glucose tolerance test (OGTT) and an intra venous glucose infusion (IIGI) will be performed.

DETAILED DESCRIPTION:
INTRODUCTION

Nonalcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease in developed countries affecting approximately 30 % of the general adult population. The disease is defined by an increased fat accumulation in the liver cells (>5 %), not caused by excessive alcohol intake (a threshold of 20 g per day for women and 30 g per day for men), autoimmunity, drugs or viral hepatitis. The histological spectrum of NAFLD ranges from simple steatosis to non-alcoholic steatohepatitis (NASH). Simple steatosis defined as steatosis without injury of the hepatocytes in form of ballooning and NASH defined as the presence of hepatic steatosis and inflammation with ballooned hepatocytes with or without fibrosis. The degree of fibrosis is an important prognostic factor and is related to liver related complications and mortality.

Diabetes is the single most important cause of end-stage renal disease (ESRD). Furthermore, more than 25 % of patients with moderate to severe chronic kidney disease (CKD) have pre-diabetic characteristics such as impaired glucose tolerance or impaired fasting glucose. NAFLD represents an important pathogenic factor in the development of type 2-diabetes and is associated with an increased risk of cardiovascular disease, insulin resistance and overweight.

Previous studies of patients with CKD with/without diabetes demonstrated, with less sensitive ultrasonic methods than what the investigators plan to use in the present project, a high prevalence of NAFLD. Furthermore, the presence of both NAFLD and CKD is likely to increase the risk for cardiovascular diseases and mortality, particular among overweight patients. NAFLD is present in both diabetic and nondiabetic patients with ESRD. The co-existence of CKD, NAFLD and gluco-metabolic disturbances, including diabetes, is a research topic with increasing focus on. Co-morbidities in CKD such as impaired insulin sensitivity, diabetes, impaired calcium-phosphate metabolism, hypertension and hypertriglyceridemia constitute risk factors for NAFLD. Unfortunately, several treatments of CKD, including kidney transplantation, have been shown to impair lipid metabolism and increase insulin resistance especially in the liver. Importantly, lifestyle changes and medical treatment modalities have been shown to have only minor impact on reducing the prevalence of these disturbances in patients with CKD.

In patients with NAFLD, either due to metabolic stress (obesity) or toxic substances (immunosuppressive treatment), liver damage and the impact on insulin resistance is reflected in characteristic modifications of metabolites and lipids in liver tissue, as well as in circulating blood, which may help to identify and interpret the pathogenesis of liver damage in the setting of CKD and transplantation. One recent hypothesis for linking liver damage and CKD involves a change in gut microbiota due to impaired renal function, leading to a leaky gut with damage of the gut-blood barrier. This transfers gut microbiota metabolites to the blood, leading to a pathogen-associated molecular pattern, reflected in changes in lipidomic and metabolomic profile in the blood. Such changes have in other conditions been associated with insulin resistance and have been linked to liver damage leading to NAFLD and later potentially fibrosis.

The role of bile acids and entero-endocrinology (including the incretin hormones glucagon like peptide 1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP)) in the development of NAFLD in CKD patients remains unknown. There are also clear limitations of the current knowledge of NAFLD and its potential role in gluco-metabolic changes and new-onset diabetes often seen after kidney transplantation. Delineation of these issues may provide new treatment targets for the benefit of patients. Risk factors for NAFLD among patients with CKD have only been investigated in small-scale studies with often inadequate methods. No studies have investigated the impact of fat lipid content measured by MR spectroscopy in kidney transplanted patients.

New therapeutic strategies for the diagnosis and management of NAFLD in patients with CKD and kidney transplanted patients with prediabetes are needed and important challenges in the elucidation of the etiology, pathogenesis and prevalence of NAFLD in CKD and transplanted patients exist. Thus, this project will bring new knowledge among a group of patients with high morbidity and an increased risk of mortality - a knowledge that may provide new guidelines for prevention and treatment of NAFLD.

Objectives

The primary objective of this project is to investigate the effect of kidney transplantation compared to healthy control persons, on the development and progression of the fat accumulation by MR spectroscopy and the monitoring of the glucometabolic, enteroendocrine, lipidomic and metabolomic profiles.

Kidney transplanted patients with previous prediabetes or normal glucose tolerance will be examined. The fat accumulation in the liver will be measured by MR spectroscopy and the prevalence of NAFLD will be investigated.

Furthermore, secondary objectives are to investigate changes in lipodomic and metabolomic related profiles, insulin secretion and sensitivity, secretion and content of bile acids, GLP-1, GIP, glucagon and amino acids before transplantation compared to after transplantation.

Data and statistical analysis

The null hypothesis is that there is no difference in relative liver fat values before and after kidney transplantation. The alternative hypothesis is that there is an increase by 50% in relative liver fat values measured by MR spectroscopy after kidney transplantation compared to pre-transplant values. In the literature a prevalence of NAFLD of 60-70% in type 2- diabetic patients defined by a liver fat content above 6% is known. With an estimated standard deviation of 15% a two-sided t-test with α=0.05 and power of 80%, a sample size of 16 patients in a paired design is needed to demonstrate a difference between the time points of 50%.

After completion of the study and data completion the results are analysed according to primary and secondary endpoints. Results are reported as mean values with confidence interval or median and range. Data are analysed with parametric (normally distributed data) or non-parametric statistics (non-normal distributed data). A 95 % confidence interval is accepted as statistically significant (p < 0.05).

All data will be pseudo anonymised.

ELIGIBILITY:
Inclusion Criteria (kidney transplanted patients):

* Outpatient at the department of nephrology at either Rigshospitalet or Herlev Hospital scheduled for a kidney transplantation with a living donor
* Impaired glucose tolerance: fasting glucose concentration < 7,0 mmol/ l and a 2-hour glucose load ≥ 7,8 mmol/ l and < 11,1 mmol/ l OR Impaired fasting glycaemia: Fasting blood glucose ≥ 6,1 mmol/ l and < 7,0 mmol/ l and a 2-hour glucose load < 7,8 mmol/ l OR Normal glucose tolerance: fasting glucose concentration < 6,1 mmol/ l and a 2-hour glucose load < 7,8 mmol/ l.

Inclusion criteria (control group):

* Normal kidney function
* Normal glucose tolerance

Exclusion Criteria:

* End stage liver disease as diagnosed by MELD (model for end stage liver disease) criteria OR
* At the waiting list for liver transplantation OR
* Daily alcohol intake above 20 g and 30 g for women and men respectively OR
* Known hepatitis A, B or C or hepatocellular carcinoma or other known liver disease OR
* Pregnancy OR
* Weight > 130 kg OR
* Implanted pacemaker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Total number of participants: 32 divided in two Groups:
  * 16 kidney transplanted patients
  * 16 healthy control persons
  The 16 kidney transplanted patients are scheduled for kidney transplantation with a living donor at Rigshospitalet. They will be recruited from the donor- and recipient register for kidney transplantation at Rigshospitalet and Herlev Hospital.
  The 16 healthy persons in the control group will be recruited through advertisement.
  All participants are screened by an OGTT before inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Changes in relative lipid signal measured by MR spectroscopy in the liver before kidney transplantation compared with three and twelve months after kidney transplantation | Kidney transplanted patients: 3 visits á 1 hour (baseline (before transplantation), three months and twelve months after transplantation), Control group: One hour
  Liver signal is measured by MR spectroscopy (the non-invasive method for determination of NAFLD)

SECONDARY OUTCOMES:
Prevalence of fibrosis in the liver before and after kidney transplantation measured by fibroscan. | Kidney transplanted patients: 3 visits x 15 minutes (baseline (before transplantation), three months and twelve months after transplantation), Control group: 15 minutes
  Measured by fibroscan of the liver (unit: kPa)
Prevalence of fibrosis in the liver before and after kidney transplantation measured in clinical index (NAFLD fibrosis score). | Kidney transplanted patients: 3 visits á one day (baseline (before transplantation), three months and twelve months after transplantation), Control group: One day
  NAFLD Fibrosis Score (consisting of age, alat, asat, Platelet Count, albumin and BMI).
Prevalence of fibrosis in the liver before and after kidney transplantation measured by clinical index (FIB-4 score). | Kidney transplanted patients: 3 visits á one day (baseline (before transplantation), three months and twelve months after transplantation), Control group: One day
  Fibrosis-4 score (consisting of age, alat, asat and Platelet Count)
Glycemic variability associated with NAFLD, as measured by MR spectroscopy, before and after kidney transplantation | Kidney transplanted patients: 4 days x3 visits (baseline (before transplantation), three months and twelve months after transplantation), Control group: 4 days
  Glycemic variability is evaluated from CGM (continuous monitoring glucose) data as standard deviation, SD.
Mean glucose associated with NAFLD, as measured by MR spectroscopy, before and after kidney transplantation | Kidney transplanted patients: 4 days x3 visits (baseline (before transplantation), three months and twelve months after transplantation), Control group: 4 days
  Values for mean glucose [mmol/ l] are evaluated from CGM (continuous monitoring glucose) data.
Change in insulin secretion during an OGTT compared with an IIGI before and at three and twelve months after transplantation and the association to NAFLD. | Kidney transplanted patients: 2 days x3 (baseline (before transplantation) and after three and twelve months after transplantation, Control group: 2 days
  Fasting levels insulin are taken before start of the test. Blood samples for measurements of insulin are taken 12 times throughout the test (time = 10 min, 15 min, 20 min, 30 min, 40 min, 50 min, 60 min, 70 min, 90 min, 120 min, 150 min, 180 min).
Change in insulin sensitivity during an OGTT compared with an IIGI before and at three and twelve months after transplantation and the association to NAFLD. | Kidney transplanted patients: 2 days x3 (baseline (before transplantation) and after three and twelve months after transplantation, Control group: 2 days
  Insulin Sensitivity Index is calculated as 10,000/ Square root of [fasting glucose X fasting insulin] [mean glucose X mean insulin during] according to Matsuda et al.
  Fasting levels of insulin and glucose are taken before start of the test. Glucose is measured every 5 minutes from time = 0 until time = 120, and every 10 minutes from time = 120 minutes to the end, time = 180 minutes.
  Blood samples for measurements of insulin are taken at time = 0 min, 10 min, 15 min, 20 min, 30 min, 40 min, 50 min, 60 min, 70 min, 90 min, 120 min, 150 min and 180 min.
The secretion and content of GLP-1 and GIP during an OGTT before and after kidney transplantation analysed from blood samples | Kidney transplanted patients: 3 hours x3 visits - through study completion (baseline (before transplantation) and after three and twelve months after transplantation, Control group: 3 hours
  Measured by blood samples during an oral glucose tolerance test. Fasting levels of GLP-1, GIP and glucagon are taken before start of the tests. Blood samples for measurements of GLP-1, GIP and glucagon are taken 12 times throughout the tests (time = 10 min, 15 min, 20 min, 30 min, 40 min, 50 min, 60 min, 70 min, 90 min, 120 min, 150 min, 180 min).
The secretion and content of GLP-1, GIP and glucagon during an IIGI before and after kidney transplantation analysed from blood samples | Kidney transplanted patients: 4 hours x3 visits - through study completion (baseline (before transplantation) and after three and twelve months after transplantation, Control group: 4 hours
  Fasting levels of GLP-1, GIP and glucagon are taken before start of the tests. Blood samples for measurements of GLP-1, GIP and glucagon are taken 12 times throughout the tests (time = 10 min, 15 min, 20 min, 30 min, 40 min, 50 min, 60 min, 70 min, 90 min, 120 min, 150 min, 180 min).
  The results from the IIGI will be compared with the results from the OGTT.
The effect of GLP-1 and GIP on insulin and glucagon response to arginine | Kidney transplanted patients: 4 hours x3 visits - through study completion (baseline (before transplantation) and after three and twelve months after transplantation, Control group: 4 hours
  Average plasma insulin and glucagon concentrations 10 minutes following arginine bolus at the end of the examination.
  Blood samples are collected at time 182, 184, 186 and 190 minutes
The secretion and content of bile acids analysed from blood samples before and after kidney transplantation and the association to NAFLD | Kidney transplanted patients: 1 day x 3 visits - through study completion (baseline (before transplantation) and after three and twelve months after transplantation, Control group: 1 day
  Measured by fasting blood samples. Blood samples will be analysed according to total and fractionated bile acids.
Change in metabolomics before kidney transplantation compared with three and twelve months after kidney transplantation, analysed from blood samples and the association with the difference in liver fat measured by MRS. | Kidney transplanted patients: 3 visits (baseline (before transplantation), three months and twelve months after transplantation), Control group: One day
  Blood samples are collected and analysed
Acute illness of non-renal or hepatic origin | Only kidney transplanted patients: Ongoing for up to 15 months - baseline until last visit (twelve months after transplantation)
  Information from Medical records.
Death rate during follow up in the Group of kidney transplanted patients | Only kidney transplanted patients: Ongoing for up to 15 months - baseline until last visit (twelve months after transplantation)
  Information from medial records.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Feldt-Rasmussen, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Nephrology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No